CLINICAL TRIAL: NCT07026591
Title: Epilepsy and Driving
Acronym: EPICO
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CSY_2025_4
Record Dates: First submitted 2025-05-27; First posted 2025-06-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- epilectic patients: Individuals with epilepsy who drive at least once a month
- healthy volunteers: healthy volunteers driving at leat once a month, matched to epileptic patients on age (+-/ 5 years), sex and driving experience (+/-3 years)

SUMMARY:
Epilepsy can lead to cognitive impairments, particularly in attention, which may affect daily activities such as driving. Driving plays a key role in maintaining autonomy and is essential for the social and professional integration of people with epilepsy. Therefore, assessing fitness to drive is a major issue for individuals with epilepsy.

French legislation governing driving for people with epilepsy clearly outlines the periods during which a person is not permitted to drive. However, the means or methods for evaluating driving fitness in these individuals are not well defined. Currently, assessment is based more on a medical consultation than on a comprehensive evaluation of driving ability.

Using a driving simulator in combination with an EEG could be a valuable approach to better assess the impact of epilepsy-related cognitive impairments on driving performance.

ELIGIBILITY:
Inclusion Criteria

* Aged between 18 and 65 years
* Holder of a category B driving license
* Active driver: drives at least once a month
* No medical condition contraindicating driving, except for epilepsy
* Provides explicit consent to participate in the study
* Affiliated with or a beneficiary of a social security scheme

Exclusion Criteria:

* Subject to legal protection (guardianship and curatorship are accepted for individuals with epilepsy, as this population represents a significant proportion of our institution's patients)
* Pregnant or breastfeeding women
* Known cybersickness (virtual reality or simulator sickness)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Epileptic patients and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Speed | Day 0
  Mean speed during the simulated driving task
Phasic alertness | Day 0
  Phasic alertness on neuropsychological test (TAP)
Lane position | Day 0
  Mean lane position during the simulated driving task
Braking time | Day 0
  Mean braking time during the simulated driving task
Information processing time | Day 0
  Mean information processing time during the simulated driving task
Sustained attention | Day 0
  Sustained attention on neuropsychological test (TAP)
Divided attention | Day 0
  Divided attention on neuropsychological test (TAP)
Visual scanning | Day 0
  Visual scanning on neuropsychological test (TAP)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut La Teppe, Tain-l'Hermitage, France